CLINICAL TRIAL: NCT06697366
Title: Liposomal Irinotecan in Combination with Sintilimab in Second-Line Treatment of Progressive Gastric Cancer, a Single-Arm, Single-Center, Open-Label, Phase II Clinical Study
Brief Title: Liposomal Irinotecan Combined with Sintilimab for Second-line Treatment of Progressive Gastric Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hao Li, Principal Investigator, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-OBU-SH-GC-Ⅱ-013
Record Dates: First submitted 2024-11-14; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; irinotecan liposome; Sintilimab; second-line treatment
MeSH Terms: conditions — Stomach Neoplasms | interventions — irinotecan sucrosofate; sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment (Experimental): The patients with Progressive Stage Gastric Cancer will be enrolled and given Sintilimab: 200 mg over 1 hour IV, given every 3 weeks. Irinotecan Liposome Injection II: 56.6 mg/m2 (free base) every 3 weeks, depending on the dose.
  Sequence of administration: Sindilizumab and Irinotecan Liposome Injection II will be given sequentially.
  Pre-treatment medication: Dexamethasone and antiemetic (or prophylactic irinotecan if preferred according to hospital practice).
  Interventions: Drug: Irinotecan liposome injection Ⅱ; Drug: Sintilimab

INTERVENTIONS:
Drug: Irinotecan liposome injection Ⅱ — 56.6 mg/m2，Q3W
Drug: Sintilimab — 200mg，Q3W

SUMMARY:
Evaluating the efficacy and safety of irinotecan liposome injection in combination with Sintilimab in the second-line treatment of progressive gastric cancer

DETAILED DESCRIPTION:
This is a single-center, open, single-arm clinical study to evaluate the efficacy and safety of irinotecan liposome injection in combination with Sintilimab in the second-line treatment of progressed gastric cancer, and to provide more clinical treatment options for gastric cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, gender is not limited;
2. Pathologically confirmed adenocarcinoma (originating from the stomach and gastroesophageal junction);
3. Clinical documentation of failure of prior standard therapy (treatment with at least 1 cycle of standard chemotherapy regimen, disease progression or intolerance during treatment, or disease progression after completion of treatment).
4. An Eastern Cooperative Oncology Group (ECOG) physical status score of 0 to 2;
5. Have equivalent organ function, i.e., meet the following criteria:

   a.Routine blood tests:
   1. Neutrophils ≥ 1.5 × 109 /L;
   2. Leukocytes ≥ 3.5 × 109 /L;
   3. Platelets ≥ 75 × 109 /L;
   4. hemoglobin ≥70 g/L; b. Biochemical examination:

   <!-- -->

   1. Total bilirubin ≤ 1.5 × upper limit of normal (ULN) (subjects with biliary obstruction, after biliary drainage ≤ 5 × ULN);
   2. ≤ 5 x ULN for alanine aminotransferase (AST) and alanine aminotransferase (ALT) in subjects with liver metastases
   3. Albumin level ≥ 28 g/L;
   4. creatinine clearance ≥ 60 ml/min; c.Cardiac function tests:

   <!-- -->

   1. normal ECG or abnormal ECG (not clinically significant in the judgment of the investigator)
   2. Left ventricular ejection fraction (LVEF) ≥ low limit of normal;
6. Previous surgery, radiotherapy, chemotherapy or other anti-tumor treatment need to end the treatment for 4 weeks or more, and the general physical condition or related adverse reactions have recovered (toxic reaction ≤ grade 1) or reached a stable state;
7. Participate voluntarily and sign the informed consent form;
8. Good compliance, agree to cooperate with the survival follow-up.

Exclusion Criteria:

1. Patients previously treated with irinotecan;
2. Subjects with ascites requiring clinical intervention (including subjects with moderate to large amounts of ascites, if the subject's ascites needs to be stabilized for more than 4 weeks after drainage);
3. Clinically significant gastrointestinal-like illness (including bleeding, infectious inflammation, perforation, obstruction, or diarrhea greater than grade 1);
4. second primary malignant tumor within 5 years (except for cured carcinoma in situ, basal or squamous cell skin cancer; subjects with other previous neoplasms that have not recurred within 5 years may be enrolled);
5. Suffering from uncontrolled cardiac or cerebral diseases or clinical symptoms, including but not limited to: ① NYHA class III or higher heart failure; ② unstable angina; ③ myocardial infarction or stroke within 6 months; ④ supraventricular or ventricular arrhythmia requiring treatment or intervention; ⑤ uncontrollable hypertension (systolic blood pressure >150 mmHg and/or diastolic blood pressure >90 mmHg after optimal treatment) ;
6. Subjects with known active hepatitis B (HBsAg positive and HBV DNA ≥ 103 copies or ≥ 1000 U/ml);
7. Active infection or unexplained fever >38.5°C during the Screening Period or on the day of dosing (in the investigator's judgment, fever due to neoplasia may be enrolled), which, in the investigator's judgment, would interfere with the subject's participation in this trial or interfere with the evaluation of efficacy;
8. Known hypersensitivity to any component of irinotecan hydrochloride liposomes or other liposomes;
9. Pregnant or lactating women;
10. Positive screening blood (urine) pregnancy test in women of childbearing potential (male and female subjects should use reliable contraception to prevent pregnancy during the trial and for 3 months after the last dose);
11. other medical or social problems that, in the judgment of the investigator, may affect the subject's ability to sign an informed consent, to participate in the trial study, or to influence the interpretation of the trial results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-11-20 (Estimated)

PRIMARY OUTCOMES:
overall response rate,ORR | up to two years
  the best response rate

SECONDARY OUTCOMES:
progression free survival,PFS | up to two years
  from first dose treatment to disease progression
Disease control rate,DCR | up to two years
  Proportion of cases with complete remission, partial remission and stabilization of lesions
adverse events, AE | up to two years
  treatment related adverse events, TRAEs

CONTACTS AND LOCATIONS:
Overall Officials: Hao Li, Principal Investigator — Ruijin Hospital

IPD SHARING:
Plan to Share IPD: No
The researchers decided not to share